CLINICAL TRIAL: NCT05293197
Title: Phase I Trial Assessing the Safety of the Repeated Ultrasound-induced Opening of the Blood-brain Barrier in Pediatric Patients With Refractory Supra-tentorial Malignant Brain Tumors Before Chemotherapy Administration
Brief Title: Safety Study of the Repeated Opening of the Blood-brain Barrier With the SonoCloud® Device to Treat Malignant Brain Tumors in Pediatric Patients
Acronym: SONOKID
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CarThera (Industry); Gustave Roussy, Cancer Campus, Grand Paris (Other); Institut Curie (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D20181321; 2021-002790-26 (EudraCT Number)
Record Dates: First submitted 2022-02-09; First posted 2022-03-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Malignant Brain Tumor; Malignant Glioma; Embryonal Tumor
Keywords: Low intensity pulsed ultrasound (LIPU); Therapeutic ultrasound; Blood-brain barrier (BBB); Malignant brain tumor; Brain cancer; Carboplatin; Children; Adolescents
MeSH Terms: conditions — Brain Neoplasms; Glioma; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SonoCloud® (Experimental): SonoCloud® : dose escalation 6 cycles of sonication
  Interventions: Device: SonoCloud® (9 transducers)

INTERVENTIONS:
Device: SonoCloud® (9 transducers) — SonoCloud®, sonication: dose escalation 6 cycles of sonication

SUMMARY:
Purpose : the aim of this study is to assess the feasibility and safety of ultrasound-induced opening of the blood-brain barrier (BBB) with the SonoCloud-9 implantable ultrasound device in pediatric patients treated for a recurrent malignant supra-tentorial brain tumor treated with carboplatin.

Study hypothesis : the blood-brain barrier can be transiently and safely opened with pulsed low intensity ultrasound immediately prior to intravenously delivered chemotherapy. The opening of the BBB with the SonoCloud-9 system will increase the tumor exposure to carboplatin and increase progression-free and overall survival in pediatric patients treated for a recurrent malignant supra-tentorial brain tumor.

DETAILED DESCRIPTION:
Malignant brain tumors are the first cause of death by cancer in children and adolescents. The dismal prognosis of malignant brain tumors is partially due to the existence of the blood brain barrier (BBB), a physiological barrier that limits the penetration of almost all molecules from the blood stream to the brain, including antineoplastic drugs.

It has been shown that the application of low intensity ultrasound on the brain in association with intravenous microbubbles leads to transient and safe opening of the BBB. Many preclinical studies have demonstrated that ultrasound-induced opening of the BBB increases the distribution of therapeutic molecules into the brain and allows tumor control and increases survival in animal models (mice, rabbits, pigs, primates).

An innovative implantable ultrasound system, the SonoCloud device, has been developed in order to repeatedly open the BBB in synchronization with chemotherapy protocols.

This intracranial and subcutaneous device is not visible and MRI compatible and allows repeatable and ambulatory treatments. Moreover, such a device allows the delivery of low intensity ultrasound in a controlled and reproductible manner.

A phase I/IIa trial has confirmed the feasibility and safety of this technique in adult patients treated for recurrent glioblastoma with carboplatin-based chemotherapy.

This study will assess the feasibility and safety of ultrasound-induced opening of the BBB with the SonoCloud device in pediatric patients treated with carboplatin chemotherapy for a recurrent supra-tentorial malignant brain tumor. The study will determine the maximum tolerated ultrasound acoustic pressure that can be used for BBB opening and the safety of the activation of 3, then 9 transducers with the SonoCloud-9® device. Patients will follow 6 months cycles of treatment. If the treatment is well tolerated, patients will be able to be treated for 6 more cycles.

The magnitude and intensity of the BBB opening, its clinical (overall survival) and radiological (progression-free survival) efficacy will be assessed as secondary endpoints. Safety of the ultrasound contrast agent SonoVue will also be evaluated in this indication in the pediatric population.

An ancillary study will assess circulating tumor DNA (ctDNA) concentrations in patients with recurrence of a supra-tentorial malignant brain tumor, at diagnosis and during repeated opening of the BBB. The study will assess the correlation between ctDNA concentrations and tumor evolution.

ELIGIBILITY:
Inclusion Criteria:

* patient aged ≥ 5 years old and < 18 years old
* patient able to receive sonications and perform MRI studies without sedation
* diagnosis of supra-tentorial primary malignant brain tumor (e.g. malignant glioma, embryonal tumor including ATRT, ependymoma)
* recurrence or progression of brain tumor after at least a first line of standard treatment (multifocal tumors and metastatic disease allowed)
* indication of treatment with carboplatin, validated in multidisciplinary meeting
* Karnofsky performance scale index (patients ≥ 16 years old) or Lansky performance status (patients < 16 years old) > 50% (a patient with a performance status score altered by a motor deficit due to tumor infiltration will be allowed to be included)
* no threat of brain herniation or uncontrolled intracranial hypertension
* corticosteroids treatment ≤ 1mg/kg/day
* neutrophils > 1.5 x 109/L
* platelets > 100 x 109/L
* total bilirubin < 1.5x upper limit of normal, AST et ALT < 2.5x upper limit of normal
* serum creatinin < 1.5x upper limit of normal for the age or creatinine clairance >70mL/min/1.73m2 (EDTA method or 24h urine)
* coagulation parameters in the normal limits for age (fibrinogen, prothrombin time and activated clotting time)
* no grade 2 or more toxicity depending on the NCI-CTCAE v5.0 criteria
* no healed wound on the scalp
* covered by health insurance
* for patients of chilbearing age (15-17 years old) : a negative pregnancy test and an efficient method of birth control
* written consent signed by the patient (if possible) and his parents or legal representatives.

Exclusion Criteria:

* weight <15kg
* significant intra-tumoral bleeding (hematoma) or ipsilateral subdural effusion
* antineoplastic treatment other than carboplatin taken at the same time or stopped since less than:

  * 6 weeks for nitrosoureas
  * 1 month for temozolomide
  * 1 month for bevacizumab
  * 5 half-lives for tyrosin kinase inhibitors
  * 3 weeks for any other chemotherapy

for the first sonication session

* radiotherapy during the last 6 weeks
* any other cancer treated during the last 5 years
* any other uncontrolled disease or active infection
* any other co-morbidity that could compromise participation to the study (in the judgement of the clinical investigator)
* any anatomical particularity (skull thickness, thin skin) that could compromise a safe implantation of the device and/or compromise the quality of the treatment (in the judgement of the clinical investigator)
* implanted defibrillator/pacemaker, neurostimulator, cochlear implant, intracerebral ferromagnetic vascular clip
* any contraindication to general anesthesia
* any contraindication to MRI or known allergy to gadolinium or other MRI contrast agent/
* any contraindication to ultrasound contrast agent:

  * allergy to the active substance or any excipient
  * acute coronary syndrome or uncontrolled ischemic heart disease
  * chronic heart failure or history of acute heart failure or heart failure grade III or IV
  * treatment with dobutamine
  * severe pulmonary arterial hypertension
  * uncontrolled systemic hypertension
  * respiratory distress syndrome
* carboplartin hypersensitivity
* treatment with phenytoin or fosphenytoin
* earlier vaccination with attenuated alive vaccine
* diminished auditory acuity ≥ grade 3 on CTCAE classification
* history of thermoregulation disorder
* impossibility of a rigorous medical follow-up due to geographic, social or mental reasons
* pregnant and lactating women
* contemporaneous treatment by anticoagulant or platelet aggregation inhibiting drugs
* contemporaneous treatment possibly toxic for the central nervous system. The following treatments are excluded if taken less than 5 half-lives before the ultrasound session (unknown toxicity in case of BBB disruption) :

  * benzodiazepine (or any sedative or hypnotique drug)
  * antihistamine
  * proconvulsant drugs
  * butyrophenone, phenothiazine, or any "conventional" antipsychotic drug
  * barbiturate
  * MAO inhibitor
  * anticholinergic
  * anticoagulant
* any contemporaneous treatment that, in the judgement of the clinical investigator, could induce brain toxicity after BBB disruption

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity directly linked to US emissions by the SonoCloud-9® (3 transducers) | Monthly up to 12 months
  Clinical evaluation (neurological deficit, intracranial hypertension, epilepsy) during acoustic pressure dose escalation, after each sonication (48h)
Dose limiting toxicity directly linked to US emissions by the SonoCloud-9®(3 transducers) | Monthly up to 12 months
  Radiological evaluation (hemorrage, ischemia, brain swelling) during acoustic pressure dose escalation, after each sonication

SECONDARY OUTCOMES:
BBB opening intensity with the SonoCloud® device | Monthly, up to 12 months
  Grading of BBB disruption using the scale previously described (Carpentier et al 2016), after each sonication
Clinical efficacy of BBB disruption by the SonoCloud® device in association with systemic chemotherapy | Month 3
  Overall Survival (OS)
Clinical efficacy of BBB disruption by the SonoCloud® device in association with systemic chemotherapy | Month 6
  Overall Survival (OS)
Radiological efficacy of BBB disruption by the SonoCloud® device in association with systemic chemotherapy | Month 3
  Progression Free Survival (PFS) using RANO Criteria
Radiological efficacy of BBB disruption by the SonoCloud® device in association with systemic chemotherapy | Month 6
  Progression Free Survival (PFS) using RANO Criteria
Allergic adverse events related to ultrasound contrast agent SonoVue® | Monthly, up to 12 months
  Allergic reactions (cutaneous eruption, oedema, respiratory failure) in relation to the use of the ultrasound contrast agent SonoVue® for BBB disruption in the pediatric population, during and after each sonication
Cardiac adverse events related to ultrasound contrast agent SonoVue® | Monthly, up to 12 months
  Cardiac reactions (thoracic pain, cardiac failure, EKG modification) in relation with the use of the ultrasound contrast agent SonoVue® for BBB disruption in the pediatric population, during and after each sonication
Feasibility of the BBB disruption technique | Monthly, up to 12 months
  Complications associated with the implantation of the SonoCloud® device : acute pain evaluation using VAS (Visual Analogue Scale) for patients >_ 7 years old or using behavioral pain scale EVENDOL for patients <7 years old, immediately after implantation
Feasibility of the BBB disruption technique | Monthly, up to 12 months
  Complications associated with the implantation of the SonoCloud® device : acute pain evaluation using VAS (Visual Analogue Scale) for patients >_ 7 years old or using behavioral pain scale EVENDOL for patients <7 years old, at day 1 after implantation
Feasibility of the BBB disruption technique | Monthly, up to 12 months
  Complications associated with the implantation of the SonoCloud® device : chronic pain evaluation using VAS (Visual Analogue Scale) for patients >_7 years old or using behavioral pain scale EVENDOL for patients <7 years old, monthly, before each new cycle of treatment
Feasibility of the BBB disruption technique | Day 1 after implantation
  Complications associated with the implantation of the SonoCloud® device using radiological examination : device position and post-operative complication (hematoma), one day after implantation
Feasibility of the BBB disruption procedure | Monthly, up to 12 months
  Assessment of complications associated with the sonications : pain evaluation using VAS (Visual Analogue Scale) for patients >_ 7 years old or using behavioral pain scale EVENDOL for patients <7 years old at needle connexion
Feasibility of the BBB disruption procedure | Monthly, up to 12 months
  Complications associated with the implantation of the SonoCloud® device : pain evaluation using VAS (Visual Analogue Scale) for patients >_ 7 years old or using behavioral pain scale EVENDOL for patients <7 years old, during sonication
Skin complications relation to the BBB disruption procedure | Monthly, up to 12 months
  Assessment of skin complications associated with sonications : eschar and/or infection, before each cycle of treatment
Feasibility of the BBB disruption procedure | Monthly, up to 12 months
  Process evaluated by the surgeon: number of tests necessary for needle connexion to the device, at each sonication
Feasibility of the BBB disruption procedure | Monthly, up to 12 months
  Process evaluated by the surgeon : duration from needle connexion to the end of sonication, at each sonication
Feasibility of the BBB disruption procedure | During surgery
  Process evaluated by the surgeon : duration for device implantation
Biodisponibility of the SonoCloud-9® device | 12 months
  Histological analysis of tissue around the device : thickness, inflammation, biocompatibility, at explantation
Assessment of SonoCLOUD- 9® device resistance | 12 months
  Physical analysis of the device, at explantation
DNA and tumor cells concentrations in blood and cerebrospinal fluid | Monthly, up to 12 months
  Evaluation of the effect of BBB disruption with the SonoCloud-9® device on the circulation of tumoral components in the blood flow, at each cycle of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin BECCARIA, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Institut Curie, Paris
  - Service de neurochirugie Pédiatrique - Hôpital Necker- Enfants Malades, Paris
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpentier A, Canney M, Vignot A, Reina V, Beccaria K, Horodyckid C, Karachi C, Leclercq D, Lafon C, Chapelon JY, Capelle L, Cornu P, Sanson M, Hoang-Xuan K, Delattre JY, Idbaih A. Clinical trial of blood-brain barrier disruption by pulsed ultrasound. Sci Transl Med. 2016 Jun 15;8(343):343re2. doi: 10.1126/scitranslmed.aaf6086. PMID 27306666
- [Background] Idbaih A, Canney M, Belin L, Desseaux C, Vignot A, Bouchoux G, Asquier N, Law-Ye B, Leclercq D, Bissery A, De Rycke Y, Trosch C, Capelle L, Sanson M, Hoang-Xuan K, Dehais C, Houillier C, Laigle-Donadey F, Mathon B, Andre A, Lafon C, Chapelon JY, Delattre JY, Carpentier A. Safety and Feasibility of Repeated and Transient Blood-Brain Barrier Disruption by Pulsed Ultrasound in Patients with Recurrent Glioblastoma. Clin Cancer Res. 2019 Jul 1;25(13):3793-3801. doi: 10.1158/1078-0432.CCR-18-3643. Epub 2019 Mar 19. PMID 30890548
- See also: more information about the SonoCloud® device and related clinical trials — http://carthera.eu/fr/